CLINICAL TRIAL: NCT02470403
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, 2-part Study Investigating the Effect of LIK066 on Body Weight in Dysglycemic (Prediabetes or Type 2 Diabetes) and Normoglycemic Patients With Elevated Body Mass Index
Brief Title: Effect of LIK066 on Body Weight in Patients With Elevated Body Mass Index
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CLIK066X2201
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: Elevated Body Mass Index
Keywords: dysglycemic, normoglycemic, prediabetes, type 2 diabetes mellitus
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2 | interventions — licogliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1: LIK066 150 mg once daily (qd) (Experimental): LIK066 150 mg qd within 15 minutes before starting lunch
  Interventions: Drug: LIK066
- Part 1: Placebo once daily (Placebo Comparator): Matching placebo tablets of LCZ696 150 mg within 15 minutes before starting lunch.
  Interventions: Drug: LIK066
- Part 2: LIK066 75 mg twice daily (bid) (Experimental): LIK066 75 mg bid before breakfast and dinner
  Interventions: Drug: Placebo
- Part 2: LIK066 50 mg three times daily (tid) (Experimental): LIK066 50 mg tid before all 3 meals;
  Interventions: Drug: Placebo
- Part 2: Placebo three times daily (Placebo Comparator): Matching placebo tablets tid before meals.
  Interventions: Drug: LIK066

INTERVENTIONS:
Drug: LIK066 — LIK066 25 mg tablets
  Arms: Part 1: LIK066 150 mg once daily (qd); Part 1: Placebo once daily; Part 2: Placebo three times daily
Drug: Placebo — Matching placebo tablets
  Arms: Part 2: LIK066 50 mg three times daily (tid); Part 2: LIK066 75 mg twice daily (bid)

SUMMARY:
A 12-week study to assess LIK066 effect on body weight in diabetics, prediabetics and normoglycemic patients with elevated body mass index (BMI)

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with stable health condition as determined by past medical history, physical examination, electrocardiogram, and laboratory tests at screening.
* Patients with dysglycemia are patients with: Fasting plasma glucose >100mg/dL (5.6 mmol/L), or HbA1c > 5.7% and < 10% at screening.
* Fasting plasma glucose ≤250mg/dL (13.9 mmol/L) at screening.
* If treated with antidiabetic medications (other than prohibited medications), patients must be on a stable dose for 12 weeks prior to randomization and maintain the dose until the end of the study.
* Subjects must have a body mass index (BMI) within the range of 35 - 50 kg/m2 at screening, with stable body weight (± 5 kg) within 3 months prior to screening

Key Exclusion Criteria:

* Pre-existing, clinically significant gastrointestinal, liver, cardiovascular, renal or other chronic medical condition which is considered serious or unstable, other than stable cardiovascular disease, treated hypertension, dyslipidemia or other stable chronic disorders
* Clinically significant GI disorder related to malabsorption or that may affect drug or glucose absorption or history of significant gastrointestinal surgery that could affect intestinal glucose absorption
* Enrollment in a diet, weight loss or exercise programs with the specific intent of losing weight, within 3 months prior to randomization, or clinical diagnosis of any eating disorder
* Pregnant or nursing (lactating) women, and women of child-bearing potential

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2016-04-04 (Actual); Study Completion 2016-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Lincoln, Nebraska, United States

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=172

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were stratified by their glycemic status (dysglycemic or normoglycemic) and randomized to LIK066 or placebo within each stratum in each part of the study.
Groups:
- Part 1: Placebo Once Daily: Matching placebo tablets of LIK066 150 mg within 15 minutes before starting lunch.
Period: Overall Study
Arm/Group | Part 1: LIK066 150 mg Once Daily (qd) | Part 1: Placebo Once Daily | Part 2: LIK066 75 mg Twice Daily (Bid) | Part 2: LIK066 50 mg Three Times Daily (Tid) | Part 2: Placebo Three Times Daily
Started | 44 | 44 | 40 | 43 | 10
Dysglycemic | 24 | 24 | 20 | 20 | 5
Normoglycemic | 20 | 20 | 20 | 23 | 5
Completed | 42 | 43 | 40 | 39 | 10
Not Completed | 2 | 1 | 0 | 4 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Subject/guardian decision | 1 | 0 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all subjects that received any study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: LIK066 150 mg Once Daily (qd) | Part 1: Placebo Once Daily | Part 2: LIK066 75 mg Twice Daily (Bid) | Part 2: LIK066 50 mg Three Times Daily (Tid) | Part 2: Placebo Three Times Daily | Total
Number analyzed (Participants) | 44 | 44 | 40 | 43 | 10 | 181
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Part 1 (44, 44, NA,NA,NA,88) | 39.0 (12.01) | 41.3 (11.07) | NA (NA) — This arm is not for Part 1 | NA (NA) — This arm is not for Part 1 | NA (NA) — This arm is not for Part 1 | 40.2 (11.54)
  Part 2 (NA, NA, 40,43,10,93) | NA (NA) — This arm is not for Part 2 | NA (NA) — This arm is not for Part 2 | 42.9 (8.96) | 39.9 (11.22) | 43.4 (12.39) | 41.6 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 26 | 26 | 26 | 8 | 105
  Male | 25 | 18 | 14 | 17 | 2 | 76

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percent Change in Body Weight From Baseline to Week 12
Description: Triplicate body weight measurements at each visit were averaged and represented body weight at that visit. Baseline was defined to be the body weight at the last visit prior to the first treatment. Baseline is Day -1 in Part 1. Percent change is calculated as [(post baseline- Baseline) /Baseline] * 100.
  A longitudinal mixed effects model for percent change in body weight was used. The model included fixed effects of treatment, time, glycemic status (a stratification factor for randomization), the treatment-by- time interaction, the treatment-by-glycemic status interaction, the time-by-glycemic status interaction, and the treatment-by-time-by-glycemic status interaction, and Baseline body weight as a covariate.
Time Frame: Baseline, Week 12 (Day 85)
Population: The pharmacodynamics (PD) analysis set included all subjects with available PD data and no protocol deviations with relevant impact on PD data. The analysis is based on all subjects with a Baseline body weight and at least one post-Baseline body weight measurement.
Measure: Least Squares Mean (80% Confidence Interval); unit: percent change
Arm/Group | Part 1: LIK066 150 mg Once Daily (qd) | Part 1: Placebo Once Daily
Number analyzed (Participants) | 44 | 43
percent change
  All subjects (n= 42, 43) | -5.51 [-6.09 to -4.93] | 0.19 [-0.39 to 0.78]
  Dysglycemic subjects (n= 22, 23) | -6.55 [-7.34 to -5.77] | 0.29 [-0.50 to 1.09]
  Normoglycemic subjects (n= 20,20) | -4.46 [-5.31 to -3.60] | 0.09 [-0.77 to 0.94]
Statistical Analysis 1: Comparison: Part 1: LIK066 150 mg Once Daily (qd) vs Part 1: Placebo Once Daily; This analysis included all subjects. The following criteria were assessed: 1. upper confidence limit of the 80% CI for treatment difference (LIK066 - placebo) was less than 0, and 2. estimated mean treatment difference was less than or equal to -5%. The first criterion addressed whether, with high certainty, there was superior weight loss in LIK066 treated group compared to placebo. The second criterion addressed whether observed mean reduction in body weight over placebo was at least 5%; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -5.70, 80% CI 2-sided [-6.52 to -4.87]
Statistical Analysis 2: Comparison: Part 1: LIK066 150 mg Once Daily (qd) vs Part 1: Placebo Once Daily; This analysis included dysglycemic subjects. The following criteria were assessed: 1. upper confidence limit of 80% CI for treatment difference was less than 0, and 2. estimated mean treatment difference was less than or equal to -5%. The first criterion addressed whether, with high certainty, there was superior weight loss in LIK066 treated group compared to placebo. The second criterion addressed whether observed mean reduction in body weight over placebo was at least 5%; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -6.85, 80% CI 2-sided [-7.96 to -5.73]
Statistical Analysis 3: Comparison: Part 1: LIK066 150 mg Once Daily (qd) vs Part 1: Placebo Once Daily; This analysis included normoglycemic subjects. The following criteria were assessed: 1. upper confidence limit of 80% CI for treatment difference was less than 0, and 2. estimated mean treatment difference was less than or equal to -5%. The first criterion addressed whether, with high certainty, there was superior weight loss in LIK066 treated group compared to placebo. The second criterion addressed whether observed mean reduction in body weight over placebo was at least 5%; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -4.55, 80% CI 2-sided [-5.76 to -3.34]

2. Primary Outcome: Part 1: Number of Patients With Any Adverse Events, Serious Adverse Events and Death
Description: This endpoint reports patients with at least one AE (any AE), serious AE and death.
Time Frame: 12 weeks
Population: The safety analysis set included all subjects that received any study drug.
Measure: Number; unit: Patients
Arm/Group | Part 1: LIK066 150 mg Once Daily (qd) | Part 1: Placebo Once Daily
Number analyzed (Participants) | 44 | 44
Patients
  With at least one AE (any AE) | 43 | 39
  Serious AE | 1 | 0
  Death | 0 | 0

3. Primary Outcome: Part 1 and Part 2: Percent Change in Body Weight From Baseline to Week 2 (Day 14)
Description: Triplicate body weight measurements at each visit were averaged and represented body weight at that visit. Baseline was defined to be the body weight at the last visit prior to the first treatment. Part 1: Baseline is defined as Day -1. Part 2: Baseline is defined as Day 1 predose.
  Percent change is calculated as [(post baseline- Baseline) /Baseline] * 100. A longitudinal mixed effects model for percent change in body weight was used.
  The longitudinal mixed effects model included fixed effects of treatment, time, glycemic status (a stratification factor for randomization), the treatment-by-time interaction, the treatment-by-glycemic status interaction, the time-by-glycemic status interaction, the treatment-by-time-by-glycemic status interaction, a random effect for study part and baseline body weight as a covariate.
Time Frame: Baseline, Week 2 (Day 14)
Population: Pharmacodynamic set. The analysis was based on all subjects with a baseline body weight and at least one post-Baseline body weight measurement. Only data from common time points in Part 1 and Part 2 were included in the analysis, i.e., Baseline and Day 14.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent change
Groups:
- Part 1 and 2 : Pooled Placebo: Placebo subjects were pooled between the 2 parts and were considered a single treatment arm for the analyses
Arm/Group | Part 1: LIK066 150 mg Once Daily (qd) | Part 2: LIK066 75 mg Twice Daily (Bid) | Part 2: LIK066 50 mg Three Times Daily (Tid) | Part 1 and 2 : Pooled Placebo
Number analyzed (Participants) | 44 | 40 | 39 | 53
Percent change | -1.17 [-2.21 to -0.12] | -1.73 [-2.75 to -0.70] | -1.71 [-2.74 to -0.69] | 0.66 [-0.46 to 1.79]
Statistical Analysis 1: Comparison: Part 1: LIK066 150 mg Once Daily (qd) vs Part 1 and 2 : Pooled Placebo; This analysis on all subjects. The following criteria were assessed: 1. upper confidence limit of 80% CI for treatment difference was less than 0, and 2. estimated mean treatment difference was less than or equal to -5%. The first criterion addressed whether, with high certainty, there was superior weight loss in LIK066 treated group compared to placebo. The second criterion addressed whether observed mean reduction in body weight over placebo was at least 5%; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.83, 80% CI 2-sided [-2.16 to -1.51]
Statistical Analysis 2: Comparison: Part 2: LIK066 75 mg Twice Daily (Bid) vs Part 1 and 2 : Pooled Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -2.39, 80% CI 2-sided [-2.94 to -1.84]
Statistical Analysis 3: Comparison: Part 2: LIK066 50 mg Three Times Daily (Tid) vs Part 1 and 2 : Pooled Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -2.38, 80% CI 2-sided [-2.93 to -1.83]

4. Primary Outcome: Part 2: Number of Patients With Any Adverse Events, Serious Adverse Events and Death
Description: This endpoint reports patients with at least one AE (any AE), serious AE and death
Time Frame: 2 weeks
Population: The safety analysis set included all subjects that received any study drug.
Measure: Number; unit: Patients
Arm/Group | Part 2: LIK066 75 mg Twice Daily (Bid) | Part 2: LIK066 50 mg Three Times Daily (Tid) | Part 2: Placebo Three Times Daily
Number analyzed (Participants) | 40 | 43 | 10
Patients
  At least one AE (Any AE) | 40 | 43 | 10
  Serious AE | 0 | 0 | 0
  Death | 0 | 0 | 0

5. Secondary Outcome: Part 2: Percent Change in Body Weight From Baseline to Week 2 (Day 14) in LIK066 Twice Daily and LIK066 Three Times Daily Arms
Description: Triplicate body weight measurements at each visit were averaged and represented body weight at that visit. Baseline was defined to be the body weight at the last visit prior to the first treatment. Baseline is defined as Day 1 predose.
  Percent change is calculated as [(post baseline- Baseline) /Baseline] * 100. A longitudinal mixed effects model for percent change in body weight was used.
  The longitudinal mixed effects model included fixed effects of treatment, time, glycemic status (a stratification factor for randomization), the treatment-by-time interaction, the treatment-by-glycemic status interaction, the time-by-glycemic status interaction, the treatment-by-time-by-glycemic status interaction, a random effect for study part and baseline body weight as a covariate.
Time Frame: Baseline, Week 2
Population: as for outcome 1
Measure: Least Squares Mean (80% Confidence Interval); unit: percent change
Arm/Group | Part 2: LIK066 75 mg Twice Daily (Bid) | Part 2: LIK066 50 mg Three Times Daily (Tid)
Number analyzed (Participants) | 40 | 43
percent change
  Dysglycemic (n= 20, 19) | -1.99 [-2.89 to -1.09] | -1.73 [-2.62 to -0.84]
  Normoglycemic (n=20, 20) | -1.46 [-2.36 to -0.57] | -1.70 [-2.60 to -0.80]

6. Secondary Outcome: Maximum Plasma Concentration of LIK066 at Steady State (Cmax ss) in Part 1 of the Study
Description: Blood samples were collected at predose, 0.5, 1, 1.5, 2, 3, 4, 6 and 24 h postdose on Day 84. Overall glycemic status represents combination of dysglycemic and normoglycemic subjects.
Time Frame: Day 84
Population: The PK analysis set included all subjects with available PK data and no protocol deviations with relevant impact on PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: LIK066 150 mg Once Daily (qd)
Number analyzed (Participants) | 40
ng/mL
  Dysglycemic (n=22) | 1230 (328)
  Normoglycemic (n=18) | 1220 (327)
  Overall (n=40) | 1230 (323)

7. Secondary Outcome: Time to Maximum Plasma Concentration of LIK066 at Steady State (Tmax, ss) in Part 1 of the Study
Description: Blood samples were collected at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6 and 24 h post-dose on Day 84. Overall glycemic status represents combination of dysglycemic and normoglycemic subjects.
Time Frame: Day 84
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: LIK066 150 mg Once Daily (qd)
Number analyzed (Participants) | 40
hour
  Dysglycemic (n=22) | 3.02 [0.517 to 4.03]
  Normoglycemic (n=18) | 4.02 [0.517 to 6.00]
  Overall (n=40) | 3.02 [0.517 to 6.00]

8. Secondary Outcome: Area Under the Plasma Concentration-time Profile to the Time of the Last Quantifiable Concentration at Steady State (AUClast, ss) of LIK066 in Part 1 of the Study
Description: Blood samples were collected at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6 and 24 h post-dose on Day 84. Overall glycemic status represents combination of dysglycemic and normoglycemic subjects. The linear trapezoidal rule was used for AUC calculation.
Time Frame: Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 1: LIK066 150 mg Once Daily (qd)
Number analyzed (Participants) | 40
hr*ng/mL
  Dysglycemic (n=22) | 11600 (3260)
  Normoglycemic (n=18) | 12800 (4860)
  Overall (n=40) | 12100 (4050)

9. Secondary Outcome: Area Under the Plasma Concentration-time Profile to the Time of Next Dosing at Steady State (AUCtau, ss) of LIK066 in Part 1 of the Study
Description: as for outcome 8
Time Frame: Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 1: LIK066 150 mg Once Daily (qd)
Number analyzed (Participants) | 40
hr*ng/mL
  Dysglycemic (n=22) | 11600 (3260)
  Normoglycemic (n=18) | 12800 (4860)
  Overall (n=40) | 12100 (4050)

10. Secondary Outcome: The Apparent Systemic Clearance at Steady State (CLss/F, ss) of LIK066 Following Extra Vascular Administration in Part 1 of the Study
Description: as for outcome 7
Time Frame: Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Liter/hour
Arm/Group | Part 1: LIK066 150 mg Once Daily (qd)
Number analyzed (Participants) | 40
Liter/hour
  Dysglycemic (n=22) | 14.1 (4.67)
  Normoglycemic (n=18) | 13.2 (4.42)
  Overall (n=40) | 13.7 (4.52)

11. Secondary Outcome: The Apparent Volume of Distribution of LIK066 During the Terminal Elimination Phase Following Extra Vascular Administration at Steady State (Vz/F, ss) in Part 1 of the Study
Description: as for outcome 7
Time Frame: Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part 1: LIK066 150 mg Once Daily (qd)
Number analyzed (Participants) | 40
Liter
  Dysglycemic (n=14) | 110 (23.8)
  Normoglycemic (n=8) | 106 (31.2)
  Overall (n=22) | 109 (26.1)

12. Secondary Outcome: Maximum Plasma Concentration of LIK066 (Cmax) in Part 2 of the Study
Description: Blood samples were collected at pre-dose, 0.5, 1, 2, 3, 4, 4.5, 5, 6, 7 and 9 h post-dose on Day 1 and 14. Overall glycemic status represents combination of dysglycemic and normoglycemic subjects. Day 14 data reports Cmax at steady state (Cmax, ss)
Time Frame: Day 1, Day 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2: LIK066 75 mg Twice Daily (Bid) | Part 2: LIK066 50 mg Three Times Daily (Tid)
Number analyzed (Participants) | 40 | 39
ng/mL
  Day 1, Dysglycemic (n= 19, 20) | 728 (274) | 513 (176)
  Day 1, Normoglycemic (n= 19, 19) | 767 (275) | 517 (223)
  Day 1, Overall (n= 38, 39) | 747 (272) | 515 (198)
  Day 14, Dysglycemic (n= 20, 19) | 1100 (361) | 716 (282)
  Day 14, Normoglycemic (n= 20, 19) | 1030 (266) | 792 (276)
  Day 14, Overall (n= 40, 38) | 1070 (315) | 754 (278)

13. Secondary Outcome: Time to Maximum Plasma Concentration of LIK066 (Tmax) in Part 2 of the Study
Description: Blood samples were collected at pre-dose, 0.5, 1, 2, 3, 4, 4.5, 5, 6, 7 and 9 h post-dose on Day 1 and 14. Overall glycemic status represents combination of dysglycemic and normoglycemic subjects. Day 14 data reports Tmax at steady state (Tmax, ss)
Time Frame: Day 1, Day 14
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | Part 2: LIK066 75 mg Twice Daily (Bid) | Part 2: LIK066 50 mg Three Times Daily (Tid)
Number analyzed (Participants) | 40 | 39
hour
  Day 1, Dysglycemic (n= 19, 20) | 1.00 (274) [0.483 to 4.53] | 1.00 (176) [0.483 to 3.98]
  Day 1, Normoglycemic (n= 19, 19) | 1.00 (275) [0.483 to 6.00] | 0.983 (223) [0.483 to 2.00]
  Day 1, Overall (n= 38, 39) | 1.00 (272) [0.483 to 6.00] | 1.00 (198) [0.483 to 3.98]
  Day 14, Dysglycemic (n= 20, 19) | 0.983 (361) [0.483 to 4.50] | 1.00 (282) [0.500 to 3.90]
  Day 14, Normoglycemic (n= 20, 19) | 1.00 (266) [0.483 to 3.00] | 0.533 (276) [0.50 to 3.92]
  Day 14, Overall (n= 40, 38) | 0.992 (315) [0.483 to 4.50] | 1.00 (278) [0.50 to 3.92]

14. Secondary Outcome: Area Under the Plasma Concentration-time Profile to the Time of the Last Quantifiable Concentration (AUClast) of LIK066 in Part 2 of the Study
Description: Blood samples were collected at pre-dose, 0.5, 1, 2, 3, 4, 4.5, 5, 6, 7 and 9 h post-dose on Day 1 and 14. Overall glycemic status represents combination of dysglycemic and normoglycemic subjects. The linear trapezoidal rule was used for AUC calculation. Day 14 data reports AUClast at steady state (AUClast, ss)
Time Frame: Day 1, Day 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 2: LIK066 75 mg Twice Daily (Bid) | Part 2: LIK066 50 mg Three Times Daily (Tid)
Number analyzed (Participants) | 40 | 39
hr*ng/mL
  Day 1, Dysglycemic (n= 19, 20) | 3160 (571) | 3910 (840)
  Day 1, Normoglycemic (n= 19, 19) | 3280 (674) | 3870 (1360)
  Day 1, Overall (n= 38, 39) | 3220 (619) | 3890 (1110)
  Day 14, Dysglycemic (n= 20, 19) | 4600 (1050) | 4740 (1200)
  Day 14, Normoglycemic (n= 20, 19) | 4300 (1160) | 4950 (1580)
  Day 14, Overall (n= 40, 38) | 4450 (1100) | 4850 (1390)

15. Secondary Outcome: Area Under the Plasma Concentration-time Profile to the Time of Next Dosing (AUCtau) of LIK066 in Part 2 of the Study
Description: Blood samples were collected at pre-dose, 0.5, 1, 2, 3, 4, 4.5, 5, 6, 7 and 9 h post-dose on Day 1 and 14. Overall glycemic status represents combination of dysglycemic and normoglycemic subjects. The linear trapezoidal rule was used for AUC calculation. Day 14 data reports AUCtau at steady state (AUCtau, ss)
Time Frame: Day 1, Day 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 2: LIK066 75 mg Twice Daily (Bid) | Part 2: LIK066 50 mg Three Times Daily (Tid)
Number analyzed (Participants) | 40 | 39
hr*ng/mL
  Day 1, Dysglycemic (n= 19, 20) | 3170 (573) | 1340 (295)
  Day 1, Normoglycemic (n= 18, 19) | 3290 (699) | 1350 (429)
  Day 1, Overall (n= 37, 39) | 3230 (632) | 1350 (362)
  Day 14, Dysglycemic (n= 20, 19) | 4620 (1060) | 1940 (600)
  Day 14, Normoglycemic (n= 20, 19) | 4310 (1160) | 2000 (586)
  Day 14, Overall (n= 40, 38) | 4470 (1100) | 1970 (586)

16. Secondary Outcome: The Apparent Systemic Clearance at Steady State (CLss/F) of LIK066 Following Extra Vascular Administration in Part 2 of the Study
Description: Blood samples were collected at pre-dose, 0.5, 1, 2, 3, 4, 4.5, 5, 6, 7 and 9 h post-dose on Day 1 and 14. Overall glycemic status represents combination of dysglycemic and normoglycemic subjects. Day 14 data reports CLss/F at steady state (CLss/F, ss)
Time Frame: Day 1, Day 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Liter/hour
Arm/Group | Part 2: LIK066 75 mg Twice Daily (Bid) | Part 2: LIK066 50 mg Three Times Daily (Tid)
Number analyzed (Participants) | 40 | 39
Liter/hour
  Day 1, Dysglycemic (n= 19, 20) | 24.3 (3.97) [0.483 to 4.53] | 39.3 (9.42) [0.483 to 3.98]
  Day 1, Normoglycemic (n= 18, 19) | 23.8 (5.28) [0.483 to 6.00] | 40.5 (12.8) [0.483 to 2.00]
  Day 1, Overall (n= 37, 39) | 24.1 (4.59) [0.483 to 6.00] | 39.9 (11.1) [0.483 to 3.98]
  Day 14, Dysglycemic (n= 20, 19) | 17.1 (4.05) [0.483 to 4.50] | 27.8 (7.35) [0.500 to 3.90]
  Day 14, Normoglycemic (n= 20, 19) | 18.5 (4.72) [0.483 to 3.00] | 27.2 (8.50) [0.50 to 3.92]
  Day 14, Overall (n= 40, 38) | 17.8 (4.40) [0.483 to 4.50] | 27.5 (7.84) [0.50 to 3.92]

17. Secondary Outcome: The Apparent Volume of Distribution of LIK066 During the Terminal Elimination Phase Following Extra Vascular Administration (Vz/F) in Part 2 of the Study
Description: Blood samples were collected at pre-dose, 0.5, 1, 2, 3, 4, 4.5, 5, 6, 7 and 9 h post-dose on Day 1 and 14. Overall glycemic status represents combination of dysglycemic and normoglycemic subjects. Day 14 data reports Vz/F at steady state (Vz/F, ss)
Time Frame: Day 1, Day 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part 2: LIK066 75 mg Twice Daily (Bid) | Part 2: LIK066 50 mg Three Times Daily (Tid)
Number analyzed (Participants) | 40 | 39
Liter
  Day 1, Dysglycemic (n= 19, 19) | 132 (51.7) [0.483 to 4.53] | 274 (224) [0.483 to 3.98]
  Day 1, Normoglycemic (n= 18, 17) | 127 (42.4) [0.483 to 6.00] | 519 (1330) [0.483 to 2.00]
  Day 1, Overall (n= 37, 36) | 130 (46.8) [0.483 to 6.00] | 390 (919) [0.483 to 3.98]
  Day 14, Dysglycemic (n= 20, 16) | 108 (52.5) [0.483 to 4.50] | 580 (1380) [0.500 to 3.90]
  Day 14, Normoglycemic (n= 20, 19) | 112 (34.1) [0.483 to 3.00] | 267 (493) [0.50 to 3.92]
  Day 14, Overall (n= 40, 35) | 110 (43.7) [0.483 to 4.50] | 410 (997) [0.50 to 3.92]

ADVERSE EVENTS:
Arm/Group | Part 1: LIK066 150 mg Once Daily (qd) | Part 1: Placebo Once Daily | Part 2: LIK066 75 mg Twice Daily (Bid) | Part 2: LIK066 50 mg Three Times Daily (Tid) | Part 2: Placebo Three Times Daily
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/44 | 0/40 | 0/43 | 0/10
Other Adverse Events (participants affected / at risk) | 43/44 | 39/44 | 40/40 | 43/43 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: LIK066 150 mg Once Daily (qd) (N=44) | Part 1: Placebo Once Daily (N=44) | Part 2: LIK066 75 mg Twice Daily (Bid) (N=40) | Part 2: LIK066 50 mg Three Times Daily (Tid) (N=43) | Part 2: Placebo Three Times Daily (N=10)
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: LIK066 150 mg Once Daily (qd) (N=44) | Part 1: Placebo Once Daily (N=44) | Part 2: LIK066 75 mg Twice Daily (Bid) (N=40) | Part 2: LIK066 50 mg Three Times Daily (Tid) (N=43) | Part 2: Placebo Three Times Daily (N=10)
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 11 | 4 | 9 | 9 | 0
Abdominal pain (Gastrointestinal disorders) | 12 | 5 | 5 | 8 | 0
Abdominal pain lower (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 40 | 11 | 40 | 42 | 8
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 6 | 4 | 4 | 4 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 10 | 8 | 6
Flatulence (Gastrointestinal disorders) | 19 | 4 | 9 | 12 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 4 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 3 | 5 | 8 | 0
Palatal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 6 | 4 | 1
Asthenia (General disorders) | 1 | 0 | 1 | 2 | 0
Chills (General disorders) | 0 | 0 | 2 | 1 | 0
Energy increased (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 4 | 0
Feeling hot (General disorders) | 2 | 1 | 1 | 2 | 0
Feeling jittery (General disorders) | 0 | 0 | 1 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 0 | 0 | 0
Medical device site dermatitis (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1
Thirst (General disorders) | 1 | 0 | 1 | 1 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Trichomoniasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 0
Fungal test positive (Investigations) | 0 | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 3 | 6 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 9 | 16 | 13 | 10 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 4 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 2 | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.